CLINICAL TRIAL: NCT01447914
Title: A Phase II Study of the c-Met Inhibitor ARQ 197 in Patients With Relapsed, or Relapsed and Refractory Multiple Myeloma
Brief Title: Tivantinib in Treating Patients With Relapsed, or Relapsed and Refractory Multiple Myeloma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2011-03470; NCI-2011-03470 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000712984; 2011-0197 (Other: M D Anderson Cancer Center); 8984 (Other: CTEP); U01CA062461 (NIH); P30CA016672 (NIH); N01CM00039 (NIH)
Record Dates: First submitted 2011-10-04; First posted 2011-10-06 (Estimated); Results first posted 2015-03-13 (Estimated); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: Refractory Multiple Myeloma
Keywords: c-Met Inhibitor ARQ-197; tivantinib; multiple myeloma; plasma cell proliferative disorder; Hypercalcemia; hematologic malignancy; plasma cell dyscrasia; cast nephropathy; amyloidosis; osteolysis; Renal insufficiency; Anemia; Bone lytic lesions; severe osteopenia; pathologic fractures; biopsy-proven plasmacytoma
MeSH Terms: conditions — Multiple Myeloma; Hypercalcemia; Hematologic Neoplasms; Paraproteinemias; Amyloidosis; Osteolysis; Renal Insufficiency; Anemia; Bone Diseases, Metabolic; Fractures, Spontaneous | interventions — ARQ 197

ARMS (1):
- ARQ 197 Treatment (Tivantinib) (Experimental): Oral Tivantinib 360 mg twice daily continuously for each day (days 1-28) of every 4-week treatment cycle (taken as three tablets of 120 mg each). Courses continue every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Tivantinib; Other: Diagnostic laboratory biomarker analysis; Other: Questionnaire administration; Procedure: Quality-of-life assessment

INTERVENTIONS:
Drug: Tivantinib — Given at a dose of 360 mg oral (PO) twice daily continuously for each day of every 4-week treatment cycle, which will be taken as three tablets of 120 mg each.
  Other Names: ARQ 197; c-Met Inhibitor ARQ 197
Other: Diagnostic laboratory biomarker analysis — Correlative studies
Other: Questionnaire administration — Ancillary studies
Procedure: Quality-of-life assessment — Ancillary studies
  Other Names: quality of life assessment

SUMMARY:
This phase II trial studies the side effects and how well tivantinib works in treating patients with relapsed, or relapsed and refractory multiple myeloma. Tivantinib may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the overall response rate of patients with relapsed, or relapsed and refractory multiple myeloma treated with the c-Met inhibitor ARQ 197 (tivantinib) as a single agent.

II. To define the toxicities of single agent ARQ 197 in a population of patients with relapsed, or relapsed and refractory multiple myeloma.

SECONDARY OBJECTIVES:

I. To obtain preliminary evidence of the durability of responses to single agent ARQ 197, including the progression free survival (PFS), the duration of response (DOR), and the time to next treatment (TTNT).

II. To correlate the activation status of the hepatocyte growth factor (HGF)/c-Met pathway in primary myeloma cells at baseline, as defined by gene expression profiling and reverse phase protein array data, with the above measures of efficacy of ARQ 197.

III. To correlate serum and marrow HGF, HGF activator (HGFA), and soluble c-Met (sc-Met) levels with the activation status of the HGF/c-Met pathway in primary myeloma cells at baseline, and with the above measures of efficacy of ARQ 197.

TERTIARY OBJECTIVES:

I. To evaluate the symptom burden of relapsed, or relapsed and refractory multiple myeloma patients undergoing therapy with single agent ARQ 197 using the M. D. Anderson Symptom Inventory (MDASI) and its multiple myeloma module (MDASI-MM) II. To evaluate the impact of therapy with single agent ARQ 197 for relapsed, or relapsed and refractory multiple myeloma on patient reported outcomes using the European Organization for Research on the Treatment of Cancer (EORTC) Quality of Life Questionnaire (QLQ) Core 30 (QLQ-C30), and the myeloma-specific module QLQ-MY20.

III. To evaluate the impact of therapy with single agent ARQ 197 for relapsed, or relapsed and refractory multiple myeloma on the ability to collect stem cells in any patients who go on to undergo subsequent stem cell mobilization.

OUTLINE:

Patients receive tivantinib orally (PO) twice daily (BID) on days 1-28. Courses continue every 28 days in the absence of disease progression or unacceptable toxicity. Patients undergo blood, urine, and bone marrow collection for gene expression profile, proteomic profiling, and other correlative studies. Patients may complete the MDASI and its MDASI-MM, the EORTC QLQ-C30, and the myeloma-specific module QLQMY20 questionnaires at baseline and periodically during study.

After completion of study treatment, patients are followed up for 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have been previously diagnosed with histologically or cytologically confirmed symptomatic multiple myeloma, which requires the presence of all three of the following International Myeloma Working Group criteria, except as noted:

  * Clonal bone marrow plasma cells >= 10%
  * A monoclonal protein in either serum or urine
  * Evidence of end-organ damage that can be attributed to the underlying plasma cell proliferative disorder (to include one of the following):

    * Hypercalcemia (corrected calcium > 2.75 mmol/L or 11.5 mg/dL)
    * Renal insufficiency attributable to myeloma (serum creatinine > 1.9 mg/dL)
    * Anemia; normochromic, normocytic with a hemoglobin value >= 2 g/dL below the lower limit of normal, or a hemoglobin or < 10 g/dL
    * Bone lytic lesions, severe osteopenia, or pathologic fractures
    * Patients with a biopsy-proven plasmacytoma and either a serum or urine monoclonal protein will also be considered to have met the diagnostic criteria for multiple myeloma in the absence of clonal marrow plasmacytosis of >= 10%
* Patients must have measurable disease, as defined by at least one of the following:

  * Serum monoclonal protein level >= 0.5 g/dL for immunoglobulin (Ig)G, IgA, or IgM disease
  * Monoclonal protein or total serum IgD >= 0.5 g/dL for IgD disease
  * Urinary M-protein excretion of >= 200 mg over a 24-hour period
  * Involved free light chain level >= 10 mg/dL, along with an abnormal free light chain ratio
* Patients must have had at least one, but not more than four prior lines of therapy for their disease, with lines of therapy being separated by the presence of documented disease progression; using this definition, treatment with induction therapy, followed by high-dose chemotherapy and autologous stem cell transplantation, and finally by maintenance therapy, would constitute one line, provided that multiple myeloma did not meet criteria for progression at any time during this period
* Patients with relapsed disease will be considered to be those who have had progression, as defined above, off of any therapy, and who completed their therapy more than 60 days prior to the finding of progression; patients with relapsed and refractory disease will be considered to be those who have had progression, as defined above, while still on their last line of therapy, or who progressed within 60 days of finishing their most recent therapy
* Patients must have completed their most recent drug therapy directed at multiple myeloma in the following time frames:

  * Chemotherapy, biological therapy, immunotherapy, or an investigational therapy at least 3 weeks prior to starting c-Met inhibitor ARQ197
  * Corticosteroids at least 3 weeks prior to starting ARQ 197, except for a dose equivalent to dexamethasone of no greater than 4 mg/day
  * Nitrosoureas, nitrogen mustards, mitomycin C, or monoclonal antibodies at least 6 weeks prior to starting ARQ 197
  * Autologous stem cell transplantation at least 12 weeks prior to starting ARQ 197
  * Allogeneic stem cell transplantation at least 24 weeks prior to starting ARQ 197, and these patients must also not have moderate to severe active acute or chronic graft-versus-host disease
* Patients must be willing and able to provide voluntary written informed consent, with the understanding that consent may be withdrawn by the subject at any time without prejudice to their future medical care
* Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1, or 2 (Karnofsky >= 60%)
* Absolute neutrophil count (ANC) >= 1,000 cells/mm^3 without growth factors within 1 week of the initiation of treatment
* Total white blood cell count (WBC) >= 2,000 cells/mm^3 without growth factors within 1 week of the initiation of treatment
* Hemoglobin >= 8 g/dL without red blood cell transfusions within 2 weeks of the initiation of treatment
* Platelet counts of >= 100,000 cells/mm^3 for patients who have bone marrow plasmacytosis of < 50%, or >= 50,000 cells/mm^3 for patients who have bone marrow plasmacytosis of >= 50%
* Total bilirubin =< 1.5 times the upper limit of the institutional normal (ULN) values
* Total aspartate aminotransferase (AST) (serum glutamic oxaloacetic acid transaminase [SGOT]) and alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 2.5 times ULN values
* Serum creatinine within the institutional normal limits OR if the creatinine is elevated, creatinine clearance (CrCl) >= 30 mL/min., as measured by a 24-hour urine collection, or estimated by the Cockcroft and Gault formula
* Patients must have evidence of adequate cardiac function, as defined by the following:

  * Absence of New York Heart Association (NYHA) class II, III, or IV congestive heart failure
  * Absence of uncontrolled angina or hypertension
  * Absence of myocardial infarction in the previous 6 months
  * Absence of clinically significant bradycardia or other uncontrolled cardiac arrhythmia defined as grade 3 or 4 according to National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE), version 4.0
* Patients who have received radiation therapy must have completed this at least 4 weeks prior to starting therapy with ARQ 197, with the following exceptions:

  * Local radiation therapy to enhance bone healing of a pathologic fracture may have been performed, as long as it was completed at least 2 weeks prior to starting ARQ 197
  * Local radiation therapy to treat post-fracture pain that is refractory to analgesics may have been performed, as long as it was completed at least 2 weeks prior to starting ARQ197
* Patients who have undergone any recent major surgery must have done so at least 4 weeks prior to starting therapy with ARQ 197, with the following exceptions:

  * Vertebroplasty and/or kyphoplasty, which must have been performed at least 1 week prior to starting ARQ 197
  * Planned elective surgery unrelated to the patient's diagnosis of multiple myeloma, such as hernia repair, may be allowed, at the discretion of the Principal Investigator, as long as it was performed at least 2 weeks prior to starting ARQ 197, and patients have recovered fully from this procedure
* Human immunodeficiency virus (HIV)-seropositive patients with acceptable organ function who meet the patient selection criteria, and who are not on combination antiretroviral therapy, and whose absolute CD4+ count is >= 400 cells per cubic millimeter of blood, will be eligible; however, HIV positive patients on combination antiretroviral therapy will be ineligible
* Male patients must agree to use an adequate method of contraception for the duration of the study since the effects of ARQ 197 on the developing human fetus are unknown; female patients must be either post- menopausal, free from menses for >= 2 years, surgically sterilized, or willing to use two adequate barrier methods of contraception to prevent pregnancy, or must agree to abstain from heterosexual activity throughout the study; female patients of childbearing potential must have a negative serum (beta-human chorionic gonadotropin [beta-HCG]) or urine pregnancy test before receiving the first dose of ARQ 197; should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately

Exclusion Criteria:

* Patients who are receiving any concurrent investigational agent with known or suspected activity against multiple myeloma, or those whose adverse events due to agents administered more than 4 weeks earlier have not recovered to a severity of grade 0 or grade 1
* Patients who have known central nervous system involvement with multiple myeloma will be excluded from this clinical trial
* Patients who have previously been treated with another agent targeting the HGF/c-Met axis, including either monoclonal antibodies to HGF or c-Met, or small molecule inhibitors of c-Met
* Patients with a known history of allergic reactions attributed to compounds of similar chemical or biologic composition to ARQ 197
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements, in the opinion of the Principal Investigator
* Pregnant or lactating women are excluded from this study
* HIV positive patients on combination antiretroviral therapy are ineligible because of the potential for pharmacokinetic interactions with ARQ 197; however, HIV seropositive patients with acceptable organ function who meet the patient selection criteria, and who are not on combination antiretroviral therapy, will be eligible
* Patients with non-secretory multiple myeloma, active plasma cell leukemia, defined as either having 20% of peripheral white blood cells comprised of CD138+ plasma cells, or an absolute plasma cell count of 2 x 10^9/L, known amyloidosis, or known POEMS syndrome (plasma cell dyscrasia with polyneuropathy, organomegaly, endocrinopathy, monoclonal protein, and skin changes)
* Patients who have required plasmapheresis and exchange less than 2 weeks prior to initiation of therapy with ARQ 197
* Patients with known active hepatitis A, B, and/or C infection
* Patients with a "currently active" second malignancy, other than non-melanoma skin cancer and carcinoma in situ of the cervix, should not be enrolled; patients are not considered to have a "currently active" malignancy if they have completed therapy for a prior malignancy, are disease free from prior malignancies for > 5 years, and are considered by their physician to be at less than 30% risk of relapse; in addition, patients with basal cell carcinoma of the skin, superficial carcinoma of the bladder, carcinoma of the prostate with a current prostate-specific antigen (PSA) value of < 0.5 ng/mL, or cervical intraepithelial neoplasia will be eligible; finally, patients who are on hormonal therapy for a history of either prostate cancer or breast cancer may enroll, provided that there has been no evidence of disease progression during the previous three years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2011-11; Primary Completion 2014-03 (Actual); Study Completion 2014-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Orlowski, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Official Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Total Recruitment Period: November 30, 2011 to August 1, 2013. All recruitment done at University of Texas (UT) MD Anderson Cancer Center.
Groups:
- Tivantinib Treatment: Oral Tivantinib 360 mg twice daily continuously for each day of every 28 day treatment cycle (taken as three tablets of 120 mg each)
Period: Overall Study
Arm/Group | Tivantinib Treatment
Started | 16
Completed | 16
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Tivantinib Treatment
Number analyzed (Participants) | 16
Age, Continuous [Mean (Full Range); unit: years] | 66.3 [49 to 76]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 13
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 13
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 16
Prior Stem Cell Transplantation (SCT) [Number; unit: participants] — Number of participants who had or did not have SCT procedures prior beginning study.
  participants
    Prior SCT | 10
    No Prior SCT | 6

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate (ORR)
Description: ORR using International Myeloma Working Group Response Criteria, achieve at least a partial response (PR) or better: Stringent Complete Response (sCR), Complete Response (CR), Very Good Partial Response (VGPR) or Partial Response (PR): CR: Negative immunofixation on serum and urine and disappearance of any soft tissue plasmacytomas and <5% plasma cells in bone marrow; sCR: CR+Normal free light chain ratio and absence of clonal cells in bone marrow by immunohistochemistry or immunofluorescence; PR: ≥50% reduction of serum M-protein and reduction in 24-hour urinary M-protein by ≥90%; VGPR: Serum and urine M-protein detectable by immunofixation but not on electrophoresis or 90% or greater reduction in serum M-protein plus urine M-protein level <100mg per 24 hour; Stable Disease (SD): Not CR, VGPR, PR or progressive disease; Progressive Disease (PD):>25% from lowest value Serum and/or Urine M-component, new lesions or soft tissue plasmacytomas, or hypercalcemia.
Time Frame: Up to 30 days
Population: Proportion of participants reported on an intent-to-treat basis.
Measure: Number; unit: participants
Arm/Group | Tivantinib Treatment
Number analyzed (Participants) | 16
participants
  Stable Disease | 4
  Progressive Disease | 7
  Not Evaluable | 5

2. Primary Outcome: Toxicities of Single Agent Tivantinib: Grade 3 Nonhematologic or Grade 4 Hematologic Toxicities According to the Common Terminology Criteria for Adverse Events (CTCAE), Version 4
Description: Toxicities with a grade 3 nonhematologic or grade 4 hematologic toxicities according to CTCAE, version 4. Grade 3 and estimated with a 95% credible interval. Summary statistics will be provided for continuous variables.
Time Frame: Up to 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Tivantinib Treatment
Number analyzed (Participants) | 16
Participants
  Non-Hematological Grade 3- Hypertension | 1
  Non Hematological Grade 3- Syncope | 2
  Non Hematological Grade 3- Pulmonari emboli | 1
  Hematological Grade 3- Neutropenia | 4
  Non Hematological Grade 3- Fatigue | 1
  Non Hematological Grade 3- Cough | 1
  Non Hematological Grade 3- Bacteremia | 1
  Non Hematological Grade 3- Anorectal Infection | 1
  Non Hematological Grade 3- Rectal Pain | 1
  Non Hematological Grade 3- Rib Pain | 1

3. Secondary Outcome: Time to Next Treatment (TTNT)
Description: Kaplan and Meier product limit methods will be used to estimate the TTNT with 95% confidence intervals.
Time Frame: From registration on trial to next treatment or death due to any cause, whichever comes first
Measure: Median (95% Confidence Interval); unit: number of months
Arm/Group | Tivantinib Treatment
Number analyzed (Participants) | 16
number of months | 4 [1 to 15]

4. Other Pre Specified Outcome: Duration of Response
Description: Kaplan and Meier product limit methods will be used to estimate the DOR with 95% confidence intervals.
Time Frame: From first observation of partial response to the time of disease progression, assessed up to 30 days
Population: No participants responded to the therapy and no analyses were done
Arm/Group | Tivantinib Treatment
Number analyzed (Participants) | 0

5. Other Pre Specified Outcome: Progression-free Survival (PFS)
Description: Kaplan and Meier product limit methods will be used to estimate the median PFS with 95% confidence intervals. Furthermore, the univariate and multivariate Cox proportional hazards regression model will be used to identify prognostic factors for PFS.
Time Frame: From start of the treatment to disease progression or death (regardless of cause of death), whichever comes first, assessed up to 30 days
Population: No participants responded to the therapy and no analyses was done.
Arm/Group | Tivantinib Treatment
Number analyzed (Participants) | 0

6. Post Hoc Outcome: Cycles of Tivantinib Treatment Administered
Description: Number of treatment cycles completed by study participants.
Time Frame: From start of participant treatment to completion or disease progression; assessed up to 16 months
Population: No participants responded to the therapy and no analyses were done
Measure: Mean (Full Range); unit: number of treatment cycles
Arm/Group | Tivantinib Treatment
Number analyzed (Participants) | 16
number of treatment cycles | 4 [1 to 15]

ADVERSE EVENTS:
Time Frame: Adverse events collected till 30 days of the last dose of the investigational agent and include all who receive any amount of study drug. Overall collection period January 2012 to February 2014.
Arm/Group | Tivantinib Treatment
Serious Adverse Events (participants affected / at risk) | 8/16
Other Adverse Events (participants affected / at risk) | 16/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tivantinib Treatment (N=16)
Bacteremia Infection (Infections and infestations) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
Hypertension (Cardiac disorders) | 1 (1)
Neutropenia (Neutrophil count decreased) (Blood and lymphatic system disorders) | 5 (9)
Pain (General disorders) | 2 (2)
Multiple pulmonary emboli (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Syncope (Cardiac disorders) | 2 (2)
Anorectal Infection (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tivantinib Treatment (N=16)
Allergic rhinitis (Immune system disorders) | 2 (2)
Alopecia (Skin and subcutaneous tissue disorders) | 2 (2)
Anemia (Blood and lymphatic system disorders) | 3 (3)
Anxiety (Nervous system disorders) | 2 (2)
Blurred vision (Eye disorders) | 2 (5)
Chills (General disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 3 (5)
Cough (Respiratory, thoracic and mediastinal disorders) | 5 (6)
Creatinine increased (Metabolism and nutrition disorders) | 1 (1)
Depression (Nervous system disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 6 (7)
Dizziness (Nervous system disorders) | 6 (8)
Dry eye (Eye disorders) | 3 (4)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 6 (9)
Edema limbs (Musculoskeletal and connective tissue disorders) | 2 (3)
Fatigue (General disorders) | 10 (14)
Fever (Infections and infestations) | 2 (2)
Flu like symptoms (Infections and infestations) | 1 (1)
Gait distrubance (Musculoskeletal and connective tissue disorders) | 1 (1)
Diverticulitis flare (Gastrointestinal disorders) | 1 (1)
Muscle Discomfort (Musculoskeletal and connective tissue disorders) | 3 (3)
Headache (Nervous system disorders) | 2 (2)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1)
Hypertension (Cardiac disorders) | 3 (3)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1)
Hypothyroidism (Endocrine disorders) | 1 (1)
Insomnia (General disorders) | 2 (2)
Memory impairment (Nervous system disorders) | 5 (5)
Diabetes (Endocrine disorders) | 1 (1) — Note: Baseline collection.
Hyperlipidemia (Cardiac disorders) | 1 (1) — Note: Baseline collection.
Myalgia (Musculoskeletal and connective tissue disorders) | 6 (9)
Nausea (Gastrointestinal disorders) | 2 (2)
Neutrophil count decreased (Blood and lymphatic system disorders) | 5 (6)
Pain (General disorders) | 7 (12)
Paresthesia (Nervous system disorders) | 1 (1)
Peripheral motor neuropathy (Nervous system disorders) | 10 (11)
Platelet count decreased (Blood and lymphatic system disorders) | 2 (2)
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 (3)
Nocturia (Renal and urinary disorders) | 6 (6)
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Sinus bradycardia (Cardiac disorders) | 3 (3)
Sinusitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Skin and subcutaneous tissue disorders (Skin and subcutaneous tissue disorders) | 2 (2)
Tinnitus (Ear and labyrinth disorders) | 1 (1)
Upper Respiratory Infection (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Urinary tract pain (Renal and urinary disorders) | 1 (1)
Watering eyes (Eye disorders) | 2 (2)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Sore Throat (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Postnasal Drip (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less